CLINICAL TRIAL: NCT07151079
Title: Evaluation of Trans Adolescent Group ThErapy for Alleviating Minority Stress (TAG TEAM): a Randomised Controlled Trial
Brief Title: TAG TEAM - Trans Adolescent Group Therapy
Acronym: TAG TEAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110355
Record Dates: First submitted 2025-08-27; First posted 2025-09-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-08

CONDITIONS: Minority Stress; Acceptability; Psychological Distress; Anxiety; Depression in Adolescence; Coping; Wellbeing; Pride; Internalised Stigma; Community Connection
Keywords: Adolescent; Trans and gender diverse; Minority stress; Wellbeing; Group Therapy; CBT
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Masking Description: The biostatistician will be masked (blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAG TEAM Intervention Arm (Experimental): In the intervention arm Trans Adolescent Group ThErapy for Alleviating Minority stress (TAG TEAM) will be delivered in groups of 8 participants (maximum) from the same stratum. Participants will be allocated to strata based on school year level (Grades 7-9 and 10-12). Participation will occur across a 5-month period for those in the intervention arm, including approximately 2-weeks for allocation to a condition, completion of the 6-week TAG TEAM program and follow-up questionnaires at 19 weeks.
  Interventions: Behavioral: Trans Adolescent Group ThErapy for Alleviating Minority stress
- Waitlist Control (No Intervention): Those randomly allocated to the waitlist control arm from the same stratum will receive TAG TEAM after waiting a total of 19 weeks.

INTERVENTIONS:
Behavioral: Trans Adolescent Group ThErapy for Alleviating Minority stress — The intervention, Trans Adolescent Group ThErapy for Alleviating Minority stress (TAG TEAM), is a group Cognitive Behavioural Therapy (CBT) program, originally developed using co-design methodology with trans and gender diverse young people. The 6 weekly, 2-hour session TAG TEAM program aims to improve mental health and wellbeing using evidence-based cognitive and behavioural strategies to target minority stressors discrimination and internalised stigma and facilitating community connection and pride. The intervention will be delivered by a psychologist facilitator and peer facilitator, who will both be trained and supervised by clinical psychologists, to groups of 8 participants from the same stratum.
  Arms: TAG TEAM Intervention Arm

SUMMARY:
This project will study the effect of the TAG TEAM group CBT program on the mental health of trans and gender diverse adolescents. TAG TEAM was co-designed by researchers and clinicians with a group of trans and gender diverse young people to help trans and gender diverse adolescents understand and cope with minority stress. Minority stress includes experiences like discrimination and rejection. TAG TEAM focuses on learning and practicing skills to support mental health and wellbeing. It also includes group discussions and activities with other trans and gender diverse young people. TAG TEAM groups are run by a psychologist and a trans peer facilitator. A trans peer facilitator is a trans and gender diverse person who is there to share their experience of being trans and to support participants in the group sessions.

DETAILED DESCRIPTION:
Trans Adolescent Group ThErapy for Alleviating Minority stress (TAG TEAM), is a group Cognitive Behavioural Therapy (CBT) program, originally developed using co-design methodology with trans and gender diverse young people. The 6 weekly, 2-hour session TAG TEAM program aims to improve mental health and wellbeing using evidence-based cognitive and behavioural strategies.

The intervention is a group CBT program, with sessions being split into distinct themes relating to minority stress and protective factors against such stress (i.e., community connectedness, discrimination and rejection, internalised stigma, and pride) and is based on core CBT principles (e.g., assigning and reviewing between-session activities, learning and practicing techniques). The sessions will include videos of trans and gender diverse adults discussing the session themes. Each session includes a 10-minute break halfway through the session.

The randomised controlled trial (RCT) will be a two-arm parallel group superiority trial where participants are randomised in a 1:1 ratio to an intervention or waitlist control arm. A mixed method design will involve quantitative analyses to evaluate the effectiveness of the intervention compared to the waitlist control.

There will also be a qualitative sub-study where participants will participate in photovoice or semi-structured interviews to evaluate their experience of the intervention. The investigators will use photovoice to investigate participants' experiences of the group CBT program and their views and perspectives on how the intervention affected their behaviour and mental health. Photovoice is a qualitative research method where participants are asked to take photos that respond to the study aims, and are then given the opportunity to describe, discuss and display the photos. The investigators will use semi-structured interviews, questionnaires and /or focus groups to explore participants, facilitators and service providers experiences of the group CBT program and their views and perspectives on how the intervention was delivered, the content and any barriers or enablers to attending and delivering the program.

A mixed method evaluation which includes questionnaires, semi-structured interviews and/or focus groups will examine the key acceptability and implementation factors from the perspective of the participants, facilitators and service providers to explore acceptability, feasibility and appropriateness of the program, fidelity, barriers and enablers to implementation and trial process data.

ELIGIBILITY:
Participants will be enrolled into the RCT only if they meet all the inclusion criteria and none of the exclusion criteria.

Inclusion Criteria:

* Identifies as trans, non-binary, or gender diverse
* Is between the ages of 12 and 17 years inclusive
* Has completed primary school at the time of enrolment into the study
* Has current psychological stress symptomology as determined by a score of moderate or above on the DASS-Y
* Provide informed consent: All participants and parent/legal guardians must be willing to give informed consent

Exclusion Criteria:

* Has current acute suicidal symptomology as determined by a combination of clinical judgement and the results of the Ask Suicide-Screening Questions (ASQ) suicide screening tool (e.g., answer yes to question 5) to determine the risk of suicide (has an active plan and/or intent to suicide) at time of screening interview
* Is actively having treatment with any other group psychological intervention at the time of enrolment into the study
* Is not proficient in English (as the group Cognitive behaviour therapy (CBT) program will be delivered in English and funds aren't available for interpreters)
* Previous participation in the feasibility trial
* Is currently enrolled in tertiary study (e.g., undergraduate university)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Transgender, non-binary and other gender diverse participants
Enrollment: 142 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Changes in level of psychological distress measured using the total score from the Depression Anxiety Stress Scales - Youth version (DASS-Y) | Measured at baseline (week 0) and 6 weeks after enrolment.
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) will be used to measure changes in psychological distress, compared to baseline, between treatment groups (intervention versus waitlist control).
  DASS-Y is a simplified version of the Depression Anxiety Stress Scales (DASS) for use with 8-17-year-olds. It is a 21-item questionnaire to assess a young person's negative emotional state in the last week, scored on a 4-point ordinal scale by severity from 0 = not true, 1 = a little true, 2 = fairly true, to 3 = very true.
  The DASS-Y total scale is composed of 3 subscales of anxiety, depression and stress. The total instrument measures depression, anxiety and stress, overall used to measure psychological distress. The total score ranges from 0 (least psychological distress) to 63 (most psychological distress). Psychological distress will be categorised into the following ordinal scale: 0-23 - Normal, 24-29 = Mild, 30-39 = Moderate, 40-46 = Severe, and 47+ = Extremely severe.

SECONDARY OUTCOMES:
Changes in level of psychological distress measured using the total score from the Depression Anxiety Stress Scales - Youth version (DASS-Y) | Measured at baseline (week 0) and 19 weeks after enrolment.
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) will be used to measure changes in psychological distress, compared to baseline, between treatment groups (intervention versus waitlist control).
  DASS-Y is a simplified version of the Depression Anxiety Stress Scales (DASS) for use with 8-17-year-olds. It is a 21-item questionnaire to assess a young person's negative emotional state in the last week, scored on a 4-point ordinal scale by severity from 0 = not true, 1 = a little true, 2 = fairly true, to 3 = very true. The DASS-Y total scale is composed of 3 subscales of anxiety, depression and stress. The total instrument measures depression, anxiety and stress, overall used to measure psychological distress.
  The total score ranges from 0 (least psychological distress) to 63 (most psychological distress). Psychological distress will be categorised into the following ordinal scale: 0-23 - Normal, 24-29 = Mild, 30-39 = Moderate, 40-46 = Severe, and 47+ = Extremely severe.
Changes in level of anxiety measured using the Anxiety subscale of the Depression Anxiety Stress Scales - Youth version (DASS-Y) | Measured at baseline (week 0), 6 weeks and 19 weeks after enrolment.
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) will be used to measure changes in anxiety, compared to baseline, between treatment groups (intervention versus waitlist control).
  DASS-Y is a simplified version of the Depression Anxiety Stress Scales (DASS) for use with 8-17-year-olds. The DASS-Y Anxiety subscale is a 7-item questionnaire to assess a young person's anxiety in the last week, scored on a 4-point ordinal scale by severity from 0 = not true, 1 = a little true, 2 = fairly true, to 3 = very true. Questions reflect both autonomous and subjective feelings of anxiety and panic for example 'I felt scared for no reason' and 'I could feel my heart beating' and 'I felt dizzy like I was going to faint'.
  The Anxiety subscale of the DASS-Y ranges from 0 (least anxiety) to 21 (most anxiety). Anxiety scores will be categorised into the following ordinal scale: 0-5 = Normal, 6-7 = Mild, 8-12 = Moderate, 13-15 = Severe, and 16+ = Extremely severe.
Changes in level of depression measured using the Depression subscale of the Depression Anxiety Stress Scales - Youth version (DASS-Y) | Measured at baseline (week 0), 6 weeks and 19 weeks.
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) will be used to measure changes in depression, compared to baseline, between treatment groups (intervention versus waitlist control).
  DASS-Y is a simplified version of the Depression Anxiety Stress Scales (DASS) for use with 8-17-year-olds. The DASS-Y Depression subscale is a 7-item questionnaire to assess a young person's anxiety in the last week, scored on a 4-point ordinal scale by severity from 0 = not true, 1 = a little true, 2 = fairly true, to 3 = very true. Questions reflect both autonomous and subjective feelings of depression for example 'I hated my life' and 'I could not help feeling sad' and 'There was nothing nice I could look forward to'.
  The Depression subscale of the DASS-Y ranges from 0 (least depression) to 21 (most depression). Depression scores will be categorised into the following ordinal scale: 0-6 = Normal, 7-8 = Mild, 9-13 = Moderate, 14-16 = Severe, and 17+ = Extremely severe.
Changes in level of Stress measured using the Stress subscale of the Depression Anxiety Stress Scales - Youth version (DASS-Y) | Measured at baseline (week 0), 6 weeks and 19 weeks.
  The Depression Anxiety Stress Scales - Youth version (DASS-Y) will be used to measure changes in Stress, compared to baseline, between treatment groups (intervention versus waitlist control).
  DASS-Y is a simplified version of the Depression Anxiety Stress Scales (DASS) for use with 8-17-year-olds. The DASS-Y Stress subscale is a 7-item questionnaire to assess a young person's anxiety in the last week, scored on a 4-point ordinal scale by severity from 0 = not true, 1 = a little true, 2 = fairly t. Questions reflect difficulty relaxing and irritability for example 'I got upset about the little things' and 'I found it difficult to relax' and 'I was easily annoyed'.
  The Stress subscale of the DASS-Y ranges from 0 (least stress) to 21 (most stress). Stress scores will be categorised into the following ordinal scale: 0-11 = Normal, 12-13 = Mild, 14-16 = Moderate, 17-18 = Severe and 19+ = Extremely severe.
Changes in Coping as measured by the Brief Coping Orientation to Problem Experienced (Brief COPE) revised questionnaire | Measured at baseline (week 0), 6 weeks and 19 weeks after enrolment.
  Changes in participants' Coping compared to baseline, between treatment groups (intervention versus waitlist control) will be measured using the active coping, self-blame, planning, positive reframing and social withdrawal subscales of the Brief Coping Orientation to Problem Experienced (Brief COPE) revised questionnaire.
  Brief COPE revised is a measure of different types of coping and has been revised for adolescents 13-24 years: questions have been simplified and an item added to each subscale to improve reliability. 18 items will be used to assess 3 forms of coping (problem-focused, avoidant and emotion-focused). This study will use 6 subscales (active coping, positive reframing, planning, social withdrawal, acceptance and self-blame).
  Responses are based on a 4-point Likert scale from 1= "I haven't been doing this at all" to 4 = "I've been doing this a lot". On each subscale, low scores indicate low use of that particular coping strategy and vice versa. There is no total score
Changes in Wellbeing as measured by the World Health Organization-Five Well-Being Index (WHO-5) | Measured at baseline (week 0), 6 weeks and 19 weeks after enrolment.
  Changes in participants' Wellbeing, compared to baseline, between treatment groups (intervention versus waitlist control) will be measured using the World Health Organization-Five Well-Being Index (WHO-5).
  The WHO-5 wellbeing index is a validated 5-item scale measuring wellbeing over the last two weeks for children 9 years and above. Questions include 'I have felt calm and relaxed' and 'My daily life has been filled with things that interest me'. Scores range from 0 = at no time and 5 = all of the time, with the total score multiplied by 4 to obtain a score out of 100 as the "best" wellbeing possible where 0 is the worst wellbeing possible.
Changes in response to the minority stressor of internalised stigma as measured by the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A) | Measured at baseline (week 0), 6 weeks and 19 weeks after enrolment.
  Changes in response to minority stressor of Internalised Stigma, compared to baseline, between treatment groups (intervention versus waitlist control) will be measured using the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A)
  Specifically, internalised stigma, community connection, and pride will be measured using the internalised stigma, community connection, and pride subscales of the GMSR-A. The 8-item Internalised Transphobia subscale will be used to measure Internalised Stigma on a 5-point scale i.e. 0-4 ordinal scale. For example, one item states, 'I resent my gender identity or expression' and responses range from 0 (strongly disagree) to 4 (strongly agree). The highest score for this subscale is 32 where a higher score indicates higher Internalised Stigma and vice versa.
Changes in response to the minority stressor of Pride in Gender as measured by the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A) | Measured at baseline, 6 weeks and 19 weeks.
  Changes in response to minority stressor of pride in gender, compared to baseline, between treatment groups (intervention versus waitlist control) will be measured using the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A)
  Specifically, internalised stigma, community connection, and pride will be measured using the internalised stigma, community connection, and pride subscales of the GMSR-A. The 8-item Pride subscale assesses internalised stigma on a 5-point scale i.e. 0-4 ordinal scale. For example, one item states 'My gender identity or expression makes me feel special and unique' and responses range from 0 (strongly disagree) to 4 (strongly agree). The highest score for this subscale is 32, where a higher score indicates higher levels of Pride and vice versa.
Changes in response to the minority stressor of Community Connectedness as measured by the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A) | Measured at baseline (week 0), 6 weeks and 19 weeks after enrolment.
  Changes in response to minority stressor of Community Connectedness, compared to baseline, between treatment groups (intervention versus waitlist control) will be measured using the Gender Minority Stress and Resilience Measure - Adolescent version (GMSR-A)
  Specifically, internalised stigma, community connection, and pride will be measured using the internalised stigma, community connection, and pride subscales of the GMSR-A. The 5-item Community Connectedness subscale assesses internalised stigma of transphobia on a 5-point scale i.e. 0-4 ordinal scale. For example, one item states 'I feel like I belong' with responses ranging from 0 (strongly disagree) to 4 (strongly agree). The highest score for this subscale is 20 where a higher score indicates higher Community Connectedness and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Cronin, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Children's Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after de-identification, upon reasonable request.
Time Frame: Beginning 6 months following analysis and article publication, the previously described data will be available while it is being actively stored by the researchers i.e., 15 years.
Access Criteria: Researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept MCRI's conditions for access.

REFERENCES:
- [Background] Chinsen A, Cronin TJ, Pace CC, Tollit MA, Pang KC. Evaluation of a codesigned group cognitive-behavioural therapy intervention for trans young people (TAG TEAM): protocol for a feasibility trial and a subsequent pilot RCT. BMJ Open. 2024 Jan 10;14(1):e076511. doi: 10.1136/bmjopen-2023-076511. PMID 38199639